CLINICAL TRIAL: NCT00845403
Title: Antigen-specific Immune Response to Hepatitis B Virus and Influenza A (H1N1 Strain) in Utero
Brief Title: Antigen-specific Immune Response to Hepatitis B Virus in Utero
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Obstetrics & Gynaecology, Associate Professor Chong Yap Seng, National University Hospital, Singapore
Other Study IDs: DSRB D/08/376
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis B
Keywords: Hepatitis B carrier
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cord Blood of HBsAg+ mothers will be collected at delivery after seeking informed consent. Mononuclear cells (T cells and monocytes) will be isolated.Purified populations of T cells will be stimulated with different mixtures of HBV peptides covering HBV proteins and experiments of ELISPOT or intracellular cytokine staining will be carried out to detect the specificty of the responsive T cell population. In addition, T cells willbe stained with HLA-tetramers specific for different HBV epitopes to directly analyze the frequency and phenotype of HBV-specific CD8+Tcells present in cord blood.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to gain an understanding of the key components of the immune response to hepatitis B present in cord blood of HBV infected mothers.

DETAILED DESCRIPTION:
Despite the development of an effective preventive HBV vaccine, the spread of HBV virus continue, particularly in Asia, where the majority of HBV infection is acquired at birth by vertical transmission from mother to baby. HBV vertical transmission has been hypothesized to cause immune tolerance to HBV and thus promoting the subsequent HBV chronicity. Such hypothesis has never been tested and nothing is known about HBV-specific adaptive immune response occurring before birth in baby born form HBV chronically infected mothers. This study aims to gain an understanding of the key components of the immune response to hepatitis B present in cord blood of HBV infected mothers. The characterization of the HBV immune response in utero will provide informations about the cause of HBV chronicity in Asian patients in the management of baby born from HBsAg+ mothers.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with HBsAg+

Exclusion Criteria:

* Pregnant women without HBsAg+

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HBsAg+ mothers are the source of possible in utero infection.Thus, the cord blood collected from these mothers after delivery would provide information about the cause of HBV chronicity in Asian patients and about the management of baby born from HBsAg+ mothers.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Anti - viral immune response in cord blood of newborn infants born to HBV+ mothers | At birth (baseline)
  Immune response was defined as activation of innate immune effectors (NK cells, monocytes) and production of TH1 cytokines IL - 2, TNF - a and IFN - g from T cells.

SECONDARY OUTCOMES:
Expression of immune genes from immune cells | At birth (baseline)
  Expression of immune gene cells was measured using Nanostring technology and epigenetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yap Seng Chong, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore